CLINICAL TRIAL: NCT06503653
Title: Creation of a Syncope Channel for Patients Admitted to the Emergency Department for Loss of Consciousness and Not Hospitalized: Etiological Predictivity (Before/After Study)
Acronym: Sync'Hope
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Dr laura Eouzan dahan, coordonator investigator, Versailles Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: P24/01_synchope
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Syncope
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prospective part (Experimental): Prospective part: Patients admitted for syncope in the emergency department, diagnosed with syncope and not hospitalized.
  Summoned within 7 to 10 days to a cardiology day hospital for examinations adapted to each patient: ECG - ETT - Holter ECG 72h - orthostatic hypotension test - post-emergency cardiology consultation - MAPA and +/- other examinations as required.
  Interventions: Diagnostic Test: syncope channel
- Retrospective part: (Active Comparator): Retrospective part: Patients with syncope discharged home from the emergency department, before the creation of the network:
  * Information sent to patients and record of patient's non-opposition;
  * Patients are called back by telephone or, failing that, by a trusted support person or attending physician;
  * What happens to these patients? Have they seen a cardiologist within 10 days? What additional examinations did they have in town? Recurrence? Did they return to the emergency department for the same reason?
  Interventions: Diagnostic Test: routine care

INTERVENTIONS:
Diagnostic Test: syncope channel — The procedures and investigations proposed for the etiological diagnosis of low-risk or "neither high nor low" syncope and included in the study are those recommended by the European Society of Cardiology.
  No additional procedures, invasive or non-invasive explorations or blood sampling not provided for as part of routine care will be offered or carried out as part of the study.
  The only change in practice for patients included in the "syncope pathway The only change in practice concerns the grouping of patients included in the "syncope pathway" into a single day at a day hospital within 10 days of their emergency consultation.
  Arms: Prospective part
Diagnostic Test: routine care — The procedures and investigations proposed for the etiological diagnosis of low-risk or "neither high nor low" syncope and included in the study are those recommended by the European Society of Cardiology.in routine care, medical examinations are carried out by specialists such as cardiologists who do not practice in hospitals
  Arms: Retrospective part:

SUMMARY:
The main aim of this study is to assess the value of creating a "syncope pathway" to optimize diagnostic performance in patients admitted to the emergency department for syncope and not hospitalized, compared with the previous pre-syncope pathway situation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over;
* Consultant at the emergency department of the Centre Hospitalier de V ersailles
* For a confirmed diagnosis:
* of recurrent syncope with low-risk criteria according to ESC 2018 (1,2) Or
* of syncope recurrent or not, not fulfilling low-risk or high-risk criteria according to the ESC 2018 definition (1,2). These patients are those with minor high-risk criteria without aggravating circumstances:

  * With no personal history of loss of consciousness whose clinical features strongly suggest syncope of rhythmic origin;
  * No structural heart disease or abnormal ECG.
* Outpatient (returning home after emergency);
* Beneficiary or beneficiary of a social security scheme (excluding AME).

Exclusion Criteria:

* Etiology of syncope identified as early as the emergency department visit;
* High-risk syncope according to ESC 2018 criteria (1,3);
* First and only episode of low-risk syncope according to ESC 2018 criteria (1,3);
* Syncope of any risk category requiring hospitalization at the discretion of the emergency physician and cardiologist;
* Legal protection by guardianship ;
* Language barrier or condition incompatible with the patient's understanding or informed adherence to the protocol;
* Opposition to the use of their pseudonymized data (for retrospective inclusions);
* Patient's refusal to give consent to participate in the study (for prospective inclusions);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-03-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
etiological diagnosis of synchope | 3 months
  Percentage of patients for whom at least one etiological diagnosis of syncope was identified.

CONTACTS AND LOCATIONS:
Locations (1):
- centre hospitalier de Versailles, Le Chesnay, Yvelines, France

IPD SHARING:
Plan to Share IPD: No